CLINICAL TRIAL: NCT04978987
Title: Identification of Disease Specific Pathways and Modifiers in Phospholamban R14del Cardiomyopathy
Acronym: DECIPHER-PLN
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 202000350 / 202000351
Record Dates: First submitted 2021-01-18; First posted 2021-07-27 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Phospholamban R14del Cardiomyopathy; Heart Failure; Cardiomyopathy, Familial
MeSH Terms: conditions — Heart Failure; Cardiomyopathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * Serum and plasma
  * Skin biopsy
  * Cardiac muscle biopsy
  * Skeletal muscle biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background

A specific mutation in phospholamban (the PLN R14del mutation), has its origin in the northern parts of the Netherlands (Figure) and causes a severe lethal dilated and/or an arrhythmogenic cardiomyopathy. A large proportion of the population of Groningen (1:1000) carries this mutation. Until now, there is no specific treatment available for patients with PLN cardiomyopathy. Patients are treated like any other type of heart failure patients, although PLN cardiomyopathy has a different etiology from "usual" heart failure. Treatment is therefore insufficient; malignant ventricular arrhythmias and end-stage heart failure at a young age are very prevalent. To develop treatment options, the investigators aim to study the following knowledge gaps:

* Pathophysiology. The clinical phenotype of PLN R14del cardiomyopathy bears characteristics of both arrhythmogenic and dilated cardiomyopathy (ACM and DCM). Using an "omics" approach of plasma, cardiac and skeletal muscle of patients and controls, the investigators aim to reveal distinct pathways affected by the mutant PLN, unique to the PLN R14del cardiomyopathy. This will be related to clinical data and mutant PLN expression levels in both cardiac and skeletal muscle biopsies. Using this extensive profiling, the investigators aim to identify disease mechanisms and provide the context for future risk stratification and disease progression monitoring.
* Penetrance. Subjects with a heterozygous PLN R14del mutation show a wide variety in phenotype. Within the same family, patients can present either with over heart failure in their 20's or completely asymptomatic until at least their 70's. So far, no modifiers have been identified. The investigators will study cardiomyocytes derived from induced pluripotent stem cells from patients who are severely affected versus family members who are unaffected but carry the mutation.
* Treatment response. The investigators have identified potential treatments, and confirmed their efficacy in in vivo models of PLN cardiomyopathy. To establish their efficacy in a human setting, the investigators will generate 3D cardiac tissues of cardiomyocytes gathered from induced pluripotent stem cells of patients affected in varying degrees and subject these tissues to the treatment.

Methods:

For the above purposes, the investigators will collect and analyze the following data/materials:

* Serum and plasma of 90 PLN R14del carriers: 30 unaffected, 30 early affected and 30 end stage.
* Skin biopsy of 20 PLN R14del carriers: 10 unaffected, 10 end stage.
* Cardiac muscle biopsy (obtained during left ventricular assist device [LVAD]/ heart transplant [HTx] surgery) of 30 patients: 10 R14del, 10 arrhythmogenic cardiomyopathy, 10 dilating cardiomyopathy.
* Skeletal muscle biopsy of 10 patients: 5 R14del, 5 non R14del family members

ELIGIBILITY:
Inclusion Criteria:

* A minimum age of 18.
* Of adequate communication.
* Informed consent is obtained.
* Genetically confirmed r14del mutation in PLN, family member or other DCM/ACM

Exclusion Criteria:

* Known allergy for local anaesthetics.
* Other subgroup specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population consists of patients with PLN R14del, end-stage ACM or DCM, and non-R14del family members of the PLN r14del patients. For this study, we will include 90 PLN R14del carriers, subdivided in 30 end-stage R14del patients, 30 early abnormal and 30 unaffected family members with the PLN R14del mutation and 10 ACM, 10 DCM and 10 PLN R14del cardiomyopathy patients undergoing LVAD or HTx surgery. Finally, we will recruit a total of 5 PLN R14del cardiomyopathy patients and 5 unaffected (non-R14del) family members for the skeletal muscle biopsy collection alone.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
The level of proteins in circulating blood and cardiac- and skeletal muscle tissue | At baseline visit
  An in-dept analyses of an extensive set of proteins assessed using large scale proteomic techniques to assess differences in individual protein levels and the total proteome of the circulating blood, cardiac tissue and skeletal muscle tissue of patients clinically differentially affected by the PLN R14del mutant protein.
The level of metabolites in circulating blood and cardiac- and skeletal muscle tissue | At baseline visit
  An in-dept analyses of an extensive set of metabolites assessed using large scale metabolomic techniques to assess differences in individual metabolite levels and the total metabolome of the circulating blood, cardiac tissue and skeletal muscle tissue of patients clinically differentially affected by the PLN R14del mutant protein
The level of mRNA in circulating blood and cardiac- and skeletal muscle tissue | At baseline visit
  An in-dept analyses of an extensive set of mRNA transcripts assessed using large scale transcriptomic techniques to assess differences in individual mRNA levels and the total transcriptome of the circulating blood, cardiac tissue and skeletal muscle tissue of patients clinically differentially affected by the PLN R14del mutant protein
The level of DNA methylation in cardiac muscle tissue | At baseline visit
  An in-dept analyses of differences in individual DNA methylation levels and patterns of cardiac tissue of patients clinically differentially affected by the PLN R14del mutant protein

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands